CLINICAL TRIAL: NCT06154720
Title: Surgical Site Infection Following Episiotomy Repair in Relation to Routine Use of Postpartum Antibiotic Prophylaxis in Low Risk Population: A Randomized Controlled Trial
Brief Title: Surgical Site Infection After Episiotomy Repair Related to Routine Use of Antibiotic Prophylaxis in Low-Risk Population
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwan Elkady, Assistant Professor, Ain Shams University
Other Study IDs: Surgical Site Infection
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Surgical Site Infection
Keywords: Episiotomy Repair
MeSH Terms: conditions — Surgical Wound Infection | interventions — Anti-Bacterial Agents; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: women who received co-amoxiclav 625gm (Megamox® film-coated tablet formed of clavulanic acid 125 mg + amoxicillin 500 mg) tab twice daily for 3 days after delivery
  Interventions: Drug: Antibiotics
- Control Group: women who did not receive antibiotics.

INTERVENTIONS:
Drug: Antibiotics — After the woman had a repaired episiotomy following uncomplicated vaginal birth at 37 weeks or greater with no indication for ongoing antibiotics in the postpartum period. The patients were randomized to receive a co-amoxiclav 625mg (study group) tabs twice daily for 3 days after delivery or no antibiotic arm (control group).
  Other Names: Augmentin 625 mg; Co-amoxicalv 625 mg
  Groups: Study Group

SUMMARY:
Bacterial infections occurring during labor, childbirth, and the puerperium may be associated with considerable maternal and perinatal morbidity and mortality. Antibiotic prophylaxis might reduce wound infection incidence after an episiotomy, particularly in situations associated with a higher risk of postpartum perineal infection, such as midline episiotomy, extension of the incision, or in settings where the baseline risk of infection after vaginal birth is high. However, available evidence is unclear concerning the role of prophylactic antibiotics in preventing infections after an episiotomy.

DETAILED DESCRIPTION:
Maternal mortality is unacceptably high worldwide, with an estimated 300,000 women dying in 2017, of which around 200,000 deaths were in sub-Saharan Africa. Maternal infection, leading to sepsis, is a leading contributor to these deaths. Yet data for the incidence and cause of maternal infection are scarce.

Several pre-existing maternal conditions may increase the risk of developing bacterial infections among women expected to have uncomplicated vaginal births. These include conditions such as malnutrition, anemia, bacterial vaginosis, and group B streptococcus infections. In addition, complications during labor and childbirth (e.g. prolonged rupture of membranes, prolonged labor, lacerations of the genital tract and retained products of conception) or provider interventions (e.g. frequent vaginal examinations, operative vaginal birth (forceps, vacuum), and episiotomy) might increase the risk of infection in the puerperium.

Episiotomy is an intended incision taken on the perineum during the second stage of labor considered for indications in which failure to perform it will result in significant perineal rupture.

Spontaneous vaginal delivery (SVD) is one which occurs when a pregnant woman goes into labor without the use of drugs or other techniques to induce labor and she delivers her baby through the vagina (birth canal) without forceps, vacuum extraction, or a cesarean section. Out of the about four million deliveries occurring in the United States each year, most of them are spontaneous vaginal deliveries.

Socioeconomic status (SES) is one of the most important factors associated with medical outcomes. When SES is low, medical care is inadequate and this has been attributed to adverse outcomes. In pregnant women, low SES can increase the risk of adverse pregnancy outcomes.

Antibiotic prophylaxis is recommended to avoid infectious complications of infection-prone obstetrical procedures, such as caesarean section, manual removal of the placenta, and repair of third- or fourth-degree perineal tears. Episiotomies are anatomically similar to a second-degree perineal laceration, involving the vaginal mucosa, connective tissue, and underlying muscles, and might not warrant the routine use of prophylactic antibiotics. However, the use of prophylactic antibiotics for episiotomies seems to vary widely. While in high-income countries there is, to our knowledge, no report on the use of prophylactic antibiotics for episiotomies, and clinical recommendations do not mention their use in the absence of infection, it seems to be very common practice in some low-income countries, where the majority of women have episiotomies and receive prophylactic antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective episiotomy.
* Gestational age 37 weeks or more

Exclusion Criteria:

* Patients with pro-longed rupture of membranes (PROM >24hrs).
* pro- longed prelabour rupture of membranes (PPROM).
* Chorioamnionitis.
* Prolonged second stage of labour (>2hrs).
* Third- or fourth-degree vaginal tears.
* Instrumental delivery like forceps or vacuum.
* Retained placenta and manual removal of placenta and post partum haemorrhage.
* Anaemic patients.
* On steroid or immunocompromised status.
* Diabetic patients

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target populations of this study were all patients who underwent episiotomy repair following uncomplicated vaginal birth at 37 weeks or greater with no indication for ongoing antibiotics in the postpartum period.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
wound infection at site of episiotomy | 6 weeks
  Follow up through a visit or telephone call a weekly until 6 weeks

SECONDARY OUTCOMES:
high temperature | 6 weeks
  body temperature of 38 degrees Celsius or higher occurring on any two occasions in the first 10 days postpartum, exclusive of the first 24 hours.
Urinary tract infection | 6 weeks
  through pus cells in urine analysis
Intrauterine infection | 6 weeks
  through offensive vaginal discharge and uterine tenderness

CONTACTS AND LOCATIONS:
Overall Officials: Marwan El-Kady, MD, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams Maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No